CLINICAL TRIAL: NCT03437499
Title: Effects of Sustained Inflation or Positive Pressure Ventilation on Release of Adrenomedullin in Preterm Infants With Respiratory Failure at Birth
Brief Title: Adrenomedullin Changes After Sustained Inflation or Positive Pressure Ventilation at Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vittore Buzzi Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 300
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Lung Injury
MeSH Terms: conditions — Lung Injury | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Pressure Ventilation (Active Comparator): Positive Pressure Ventilation ( peak pressure set at 25 cmH20 and PEEP set at 5 cmH2O, with 40 inflations per minute)
  Interventions: Procedure: Positive Pressure Ventilation
- Sustained Inflation (Experimental): Prolonged inflation ( 25 cmH20 for 15 seconds) followed by PEEP set at 5 cmH2O
  Interventions: Procedure: Sustained Inflation

INTERVENTIONS:
Procedure: Sustained Inflation — Application of positive pressure by face mask with T-piece resuscitator for a prolonged period of 15 seconds at a peak pressure of 25 cmH20 followed by PEEP set at 5 cmH2O
  Arms: Sustained Inflation
Procedure: Positive Pressure Ventilation — Application of positive pressure by face mask with T-piece resuscitator at a peak pressure of 25 cmH20, PEEP set at 5 cmH2, for 40 inflations/minute
  Arms: Positive Pressure Ventilation

SUMMARY:
In this clinical trial the Investigators aimed to assess the Adrenomedullin (AM) release in urine and plasma in preterm infants undergoing Sustained Inflation or Positive Pressure Ventilation at birth to manage respiratory failure.

DETAILED DESCRIPTION:
Background and objectives: The respiratory management in the DR may play an important role in the development and prevention of lung injury. The sustained lung inflation (SI) is a promising approach to facilitate cardio-respiratory transition, but currently, although it has been shown to decrease the duration of MV, seems not to guarantee relevant benefits compared to Positive Pressure Ventilation (PPV). In order to clarify the impact of these two different approaches on lung tissues, this study measures Adrenomedullin (AM), which is a biomarker involved in lung development.

Methods: we conducted a prospective case control-study in a cohort of very low birth weight (VLBW) infants (< 1500 g) of 28+0-30+6 weeks of gestational age (GA), who received SI or PPV during stabilization in DR.

Exclusion criteria were major malformations (i.e. congenital heart disease, cerebral, lung and abdominal malformations), fetal hydrops, lack of parental consent and need for endotracheal intubation at birth.

Blood samples for AM measurement were collected at birth from the arterial umbilical cord before resuscitation maneuvers, then at 1 hour from birth and at 24 hours from birth. Moreover, urine samples were collected, in correspondence with the first urine emission while in NICU and at 24 hours of life.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 28+0 and 30+6
* need for respiratory support in the delivery room

Exclusion Criteria:

* major malformations (i.e. congenital heart disease, cerebral, lung and abdominal malformations)
* fetal hydrops
* lack of parental consent.
* Need for endotracheal intubation at birth

Ages: 28 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
AM levels in plasma and urine in preterm infants with respiratory failure | 24 hours
  to investigate, in a cohort of preterm infants with respiratory failure at birth, the short-term AM release (plasma and urine samples at different time-points) after initial resuscitation with SI or PPV.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Lista, MD PhD, Study Chair — NICU-ASST-FBF-Sacco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lista G, Boni L, Scopesi F, Mosca F, Trevisanuto D, Messner H, Vento G, Magaldi R, Del Vecchio A, Agosti M, Gizzi C, Sandri F, Biban P, Bellettato M, Gazzolo D, Boldrini A, Dani C; SLI Trial Investigators. Sustained lung inflation at birth for preterm infants: a randomized clinical trial. Pediatrics. 2015 Feb;135(2):e457-64. doi: 10.1542/peds.2014-1692. PMID 25624390
- [Result] Kitamura K, Kangawa K, Kawamoto M, Ichiki Y, Nakamura S, Matsuo H, Eto T. Adrenomedullin: a novel hypotensive peptide isolated from human pheochromocytoma. Biochem Biophys Res Commun. 1993 Apr 30;192(2):553-60. doi: 10.1006/bbrc.1993.1451. PMID 8387282
- [Result] Zhang S, Patel A, Moorthy B, Shivanna B. Adrenomedullin deficiency potentiates hyperoxic injury in fetal human pulmonary microvascular endothelial cells. Biochem Biophys Res Commun. 2015 Sep 4;464(4):1048-1053. doi: 10.1016/j.bbrc.2015.07.067. Epub 2015 Jul 18. PMID 26196743